CLINICAL TRIAL: NCT04527588
Title: Italian Translation and Cross-cultural Adaptation of the Michigan Hand Outcomes Questionnaire
Brief Title: Italian Translation of the Michigan Hand Outcomes Questionnaire
Status: Withdrawn | Type: Observational
Why Stopped: same study was published from another group
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Maurizio Calcagni, MD, University of Zurich
Other Study IDs: Michigan2020.USZ
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Hand Fracture; Hand Osteoarthritis; Hand Injury Wrist; Hand Sprain; Wrist Injuries; Wrist Fracture; Wrist Arthritis
MeSH Terms: conditions — Wrist Injuries; Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionaire Michigan — Patient-Reported Outcome Measures (PROMs) are important clinical items for evaluating injuries and recovery of the hand. The Michigan Hand Questionnaire is one of the most important.

SUMMARY:
Patient-Reported Outcome Measures (PROMs) are important clinical items for evaluating injuries and recovery of the hand. Some of the most used Questionnaires, unfortunately, are not available in Italian.

DETAILED DESCRIPTION:
Patient-Reported Outcome Measures (PROMs) are important clinical items for evaluating injuries and recovery of the hand. Some of the most used Questionnaires, unfortunately, are not available in Italian. This poses a problem when evaluating Italian speaking patients. Our aim is to develop a culturally adapted Italian version of the Michigan Hand Questionnaire. There is no risk involved for the patients, as the task of the recruited patients is to answer a survey (online and in clinics).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* native Italian speakers
* wrist/hand pathology
* trauma (fractures, tendon injuries, etc.)
* chronic pathology, the pathology has been present for at least 1 month (tenosynovitis, chronic arthrosis pain, rheumatic hand or wrist disorders)
* in case of hand/wrist surgery: at least 4 weeks have elapsed since surgery to avoid that the patient could not perform certain actions evaluated by the scale, for example lifting a pan or shopping bags, due to normal post-operative precautions.
* full possession of mental capacity

Exclusion Criteria:

* age < 18 years
* non-native Italian speakers of Italian, thus also excluding second generation Swiss Italians ("secundo")
* mental incapacity
* upper limb in cast/locked by splint (criterion in Chung's article 98) at the time of the evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Native Italian speaking patients followed by the Hand Therapy of the University Hospital Zürich and the Handtherapy Fairplay center of Bologna, IT, with a pathology of the hand/s and or wrist/s.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Validity | 3 months
  Validity will be assessed as structural validity, i.e., "the degree to which the scores of the Health-Related Patient Reported Outcome (HR-PRO) are an adequate reflection of the dimensionality of the construct to be measured" (Mokkink et al., 2010).

SECONDARY OUTCOMES:
Reliability | 3 months
  Reliability will be assessed as internal consistency (i.e., "the degree of the interrelatedness among the items" [Mokkink et al., 2010]), test-retest reliability (i.e., "the proportion of the total variance in the measurements which is due to 'true' differences between patients" [Mokkink et al., 2010]), and measurement error (i.e., "the systematic and random error of a patient's score that is not attributed to true changes in the construct to be measured" [Mokkink et al., 2010]).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, MD, Study Director — University Hospital, Zürich

IPD SHARING:
Plan to Share IPD: No
Patient-Reported Outcome Measures (PROMs) are important clinical items for evaluating injuries and recovery of the hand. Some of the most used Questionnaires, unfortunately, are not available in Italian. This poses a problem when evaluating Italian speaking patients. Our aim is to develop a culturally adapted Italian version of the Michigan Hand Questionnaire. There is no risk involved for the patients, as the task of the recruited patients is to answer a survey (online and in clinics).